CLINICAL TRIAL: NCT01519154
Title: Untersuchung Unterschiedlicher Sedationstechniken für Elektive Magnetresonanztomographie (MRT)-Diagnostik Bei Kindern Anhand Klinischer Und MRT-basierter Outcomeparameter (Propofol Versus Propofol-Ketamin)
Brief Title: Sedation MRI - Propofol Versus Propofol-Ketamin in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achim Schmitz (Other)
Responsible Party: Sponsor-Investigator, Achim Schmitz, Principal Investigator, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KEK-ZH Nr. 2011-0190; 2011DR3171 (Other: Swissmedic Referenznummer)
Record Dates: First submitted 2012-01-17; First posted 2012-01-26 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sedation
Keywords: deep sedation; propofol; ketamine; child; preschool child; infant; recovery and quality of sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Propofol 10 mg/h as maintenance infusion
  Interventions: Drug: Propofol
- Ketamine-Propofol (Experimental): Additional Ketamine at induction, Propofol 5 mg/h as maintenance infusion
  Interventions: Drug: Ketamine-Propofol

INTERVENTIONS:
Drug: Propofol — Only Propofol titrated for induction, followed by Propofol 10 mg/h as maintenance infusion
  Arms: Propofol
Drug: Ketamine-Propofol — Propofol titrated plus additional Ketamine 1 mg/kg at induction, followed by Propofol 10 mg/h as maintenance infusion
  Arms: Ketamine-Propofol

SUMMARY:
Children < 10 years of age often need deep sedation or anaesthesia to allow elective diagnostic magnetic resonance imaging; standard routine protocols are

1. propofol induction without other sedative (Propofol much as needed) or hypnotic drugs and propofol infusion 10 mg/kg h
2. propofol induction with ketamine 1 mg /kg (little repetitive Propofol doses as needed) and propofol infusion 5 mg / kg h

both protocols are compared with regard to clinical outcome and, in cases with cerebral MRI, cerebral perfusion/blood flow.

Hypothesis:

1. reduces recovery time compared to propofol mono sedation
2. combination of ketamine-propofol increases incidence of Postoperative nausea and vomiting (PONV) compared to propofol mono sedation
3. combination of ketamine-propofol increases global cerebral blood flow and changes regional distribution of cerebral perfusion compared to propofol mono sedation

ELIGIBILITY:
Inclusion Criteria:

* MRT in deep sedation
* outpatient
* > 3 months to <= 10 years

Exclusion Criteria:

* tracheal intubation required
* contraindication of ketamine or propofol
* additional painful procedure requiring analgesics

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Recovery time | 1 - 3 hours post anaesthesia
  Time from end of MRI until recovery defined as Aldrete Score = 10

SECONDARY OUTCOMES:
Demission time | 1 - 4 hours post anaesthesia
  time until demission
PONV | 24 hours
  Postoperative nausea or vomiting
Cerebral perfusion | first 10 minutes of MRI
  noninvasive measurement of cerebral perfusion by means of MRI only in patients scheduled for cerebral MRI
Incidence of emergence delirium | 1 - 4 hours post anaesthesia
Quality of sedation | during MRI, on the average 45 minutes
  Extra Propofol doses and total amount of Propofol required, movement artefacts
respiratory and cardiovascular adverse events | during sedation, on the average 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Schmitz, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland